CLINICAL TRIAL: NCT07182032
Title: Ketamine Use in Central Sensitization: a Study Evaluating the Use of Ketamine in Centrally Sensitized Endometriosis Patients
Brief Title: Ketamine in Central Sensitization
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Adi Cosic, Physician, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY20250700
Record Dates: First submitted 2025-09-16; First posted 2025-09-19 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Endometriosis; Chronic Pelvic Pain
Keywords: ketamine; central sensitization
MeSH Terms: conditions — Endometriosis | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): standard general anesthesia without ketamine
- Ketamine (Experimental): standard general anesthesia with ketamine
  Interventions: Drug: ketamine

INTERVENTIONS:
Drug: ketamine — Participants will receive general anesthesia with protocoled ketamine infusion
  Arms: Ketamine

SUMMARY:
The purpose of this research study is to see if ketamine infusion during surgery can decrease pain after surgery. Ketamine is a medication commonly used as part of anesthesia during surgery and is approved by the US FDA.

Patients will be randomized to either receive standard anesthesia with OR without ketamine. The surgical procedure will be the same regardless of which group patients are randomized to. After surgery, patients will be asked to rate their pain in the post-operative observation unit and at their two-week post-operative visit. No additional visits are required for participation in this study. The investigators estimate the surveys will take approximately 10 minutes to complete.

ELIGIBILITY:
Inclusion Criteria:

* age range 18-89
* ASA classification I-III
* outpatient elective laparoscopy for endometriosis

Exclusion Criteria:

* known allergy or contraindication to ketamine
* History of substance use disorder, including alcohol or marijuana use, both current and remote
* History of severe psychiatric illness, including schizoaffective disorder, bipolar disorder, psychosis, or decompensated psychiatric condition , excluding anxiety and depression
* Current Intraoperative complications

Ages: 18 Years to 89 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
change in pain as measured by visual analog scale | approximately post-operative day 0 and 14
  A Visual Analog Scale (VAS) is a tool for patients to rate their pain on a 100mm line, where "no pain" is at one end and "worst pain imaginable" is at the other.

SECONDARY OUTCOMES:
Intraoperative opioid consumption as measured by anesthesia charting | Intraoperatively up to 8 hours
  Reported in morphine equivalents
change in postoperative pain scores measured by numerical rating scale | approximately postoperative day 0 and 14
  NRS is a simple and widely used pain assessment tool that asks patients to rate their pain intensity on a scale from 0 (no pain) to 10 (severe pain).
incidence of postoperative nausea/vomiting as measured by patient report | postoperative day 0
change in total analgesic consumption post-surgery as measured by chart review and patient report | approximately postoperative day 0, 1 and 14
  measured in morphine milliequivalents
incidence of postoperative delirium as measured by chart review | postoperative day 0
change in central sensitization as measured by central sensitization inventory (CSI) score | approximately postoperative day 0 and 14
  The CSI consists of 25 questions, each rated on a 0-4 scale (0 = never, 4 = always). The total score ranges from 0 to 100. Higher scores indicate a greater degree of central sensitization.

CONTACTS AND LOCATIONS:
Overall Officials: Adi Cosic, DO, Principal Investigator — University Hospitals; Morgan Cheeks, MD, Principal Investigator — University Hosptials
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No